CLINICAL TRIAL: NCT06838403
Title: Effect of Masgutova Neurosensorimotor Reflex Integration on Oro-Motor Functional Skills in Children With Cerebral
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hibatuallah ehab, hebatuallah, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OME and Masgutova method
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Oro-motor; MNRI; CP (Cerebral Palsy); OME; Masgutova Method
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): Each child in the study group will receive OME program in addition to 15 minutes MNRI technique for three times per week for 6 weeks
  Interventions: Other: Oro motor excercise to study arms and controoled arms
- controlled arm (Other): Each child in both groups will receive OME program for 30 minutes three times per week for 6 months.
  Interventions: Other: Oro motor excercise to study arms and controoled arms

INTERVENTIONS:
Other: Oro motor excercise to study arms and controoled arms — Each child in both groups will receive OME program for 30 minutes three times per week for 6 months.

SUMMARY:
Cerebral palsy (CP) is a disorder of movement and/or posture caused by a non-progressive brain lesion that persists through the lifespan and has a prevalence of more than 2 per 1000 live births (Oskoui et al., 2013). It comprises a heterogeneous group of impairments that may also affect the oral motor functions needed for eating, drinking, swallowing, and articulation (Romano et al., 2017). Dysphagia is a swallowing problem that can influence the safety and efficiency of feeding. This may lead to inadequate nutritional status due to prolonged feeding times (Mishra et al., 2018), stress during mealtimes for the caregiver and/or the child, and impaired growth (Cousino and Hazen, 2013; Stevenson et al, 2006). Estimates of the prevalence of dysphagia in children with CP vary widely due to the different definitions and tools used, variability in severity of CP, and motor type. The prevalence ranges from 21% in a group of 1357 children with CP (Parkes et al., 2010), to 99% in a group of 166 severely affected children with intellectual impairment (Calis et al., 2008). Children with CP commonly have feeding disorders and dysphagia that in many instances place them at risk for aspiration with oral feeding, with potential pulmonary consequences. They also commonly have reduced nutrition/ hydration status and prolonged stressful mealtimes. The specific nature and severity of the swallowing problems may differ, at least to some degree, in relation to sensorimotor impairment, gross and fine motor limitations, and cognitive/ communication deficits. Children with generalized severe motor impairment (for 2

example, spastic quadriplegia) are likely to experience greater swallowing deficits (Calis et al., 2008; Parkes et al., 2010). Oropharyngeal dysphagia may be characterized by problems in any or all phases of swallowing (Arvedson et al., 2019). The oral cavity and pharynx are anatomically separate but functionally integrated, the two regions are involved in complex motor responses that include feeding, chewing, swallowing, speech, and respiration. The multiple sensory receptors that innervate these two regions provide the first link in reflexes that control muscles of the entire head, upper gastrointestinal tract, and airway. Most of the reflexes affect the diversity of muscles that compose the tongue, which is vital to all stages of feeding, and which continually affects the patency of the airway (Miller, 2002). The types of oral and pharyngeal problems that children with CP have include reduced lip closure, poor tongue function, tongue thrust, exaggerated bite reflex, tactile hypersensitivity, delayed swallow initiation, reduced pharyngeal motility and drooling. Impaired oral sensorimotor function can result in drooling that in turn results in impaired hydration (Santos et al., 2012). The Schedule for Oral Motor Assessment (SOMA) is an assessment tool developed for the objective assessment of oral motor function in infants, with proven reliability and validity clinical setting. The SOMA is an assessment tool designed for the objective evaluation of oral-motor functions in children, with proven reliability and validity in infants aged 8-24 months. For the 5 types of test diet, based on the cutting score after assessment in each category, subjects are classified into normal or abnormal oral-motor function groups (Reilly et al., 1995). Oral motor rehabilitation therapy in children with CP aims at reducing or eliminating swallowing disorders and promoting functional feeding (Novak et al., 2020). Some studies suggest that intervention with oral motor therapy (OMT) or oro-motor exercise (OME) has a beneficial effect on functional independence levels and improves the quality of life of patients with feeding and swallowing 3 disorder (FSD) (Sığan et al., 2013; Howe and Wang, 2013). The Masgutova Neurosensorimotor reflex integration (MNRI) Facial Reflex Integration course is directed to the specific primary reaction of facial reflexes and their integration with whole movement development and learning. It arises from the basic Neurosensorimotor Reflex Integration concept that addresses the enhancement of learning through developing movement

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effect of MNRI on:

1. Oro-motor functional skills with different food textures in children with cerebral palsy
2. Feeding level
3. Drooling

ELIGIBILITY:
Inclusion Criteria:1. Children with spastic CP both sexes 2. Both sexes 3. Age ranged from 1 to 3years and 9 months. 4. Having oromotor dysfunction and drooling. 5. Having dysphagia ranging from level 4 to 6 on FOIS. -

Exclusion Criteria:

- 1. Congenital problems of mouth and soft plate. 2. Any surgical intervention of head or mouth.

3. Gum Disorders (e.g. gingivitis). 4. Epilepsy.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Schedual for oromotor Assessment ( SOMA ) | baseline
  The SOMA is divided into four main components:
  * Oral motor challenge categories
  * Functional areas
  * Functional units
  * Discrete oral motor behaviors. Oral motor challenge categories (OMC) refer to the graded textures presented to the infant. There are seven OMC categories:
    1. Puree.
    2. Semi-solids.
    3. Solids.
    4. Bottle.
    5. Trainer cup.
    6. Cup.
    7. Crackers.
The Drooling Severity and Frequency Scale (DSFS) is a semi-quantitative assessment of the amount of drooling. It originally was developed to measure frequency and severity of drooling in individuals with cerebral palsy. Subsequently, it has been used in | baseline
  he DSFS consists of 2 questions. The first question rates severity on a five-point (1-5) scale (never drools, mild, moderate, severe, or profuse). The second question rates drooling on a four-point (1-4) scale (no drooling, occasional, frequent, or constant). The Drooling Score equals the sum of the Severity and Frequency sub-scores (range 2-9).

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided